CLINICAL TRIAL: NCT03629119
Title: PsylliumRx: Use of Dietary Fiber in Severely Obese Children to Delay the Onset of Obesity-related Health Conditions - Pilot
Brief Title: PsylliumRx Dietary Fiber Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was put on hold in March 2020 due to COVID
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ChOBFiber-P
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Childhood Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dietary Fiber Supplement (Experimental): Participants will be instructed to consume 1 tea spoon of psyllium per day for 3 months and otherwise maintain their habitual diet.
  Interventions: Dietary Supplement: Dietary Fiber Supplement

INTERVENTIONS:
Dietary Supplement: Dietary Fiber Supplement — Participants will be instructed to consume 1 tea spoon of psyllium per day for 3 months and otherwise maintain their habitual diet. Participants will be asked to keep a diary assessing bowel movement and intestinal symptoms such as bloating and flatulence beginning two weeks prior to the intervention.

SUMMARY:
The purpose of this pilot study is to assess the feasibility of a 3-month dietary fiber intervention: 1) engaging adolescents in regularly consuming a dietary fiber preparation (psyllium powder) and obtaining their parents' support, 2) recruit into a clinical pilot trial with liquid meal challenge test to study the metabolic effects of the dietary fiber preparation. A study modification will be submitted to add additional study arms for feasibility (strength training, coaching).

DETAILED DESCRIPTION:
For this 3-month clinical pilot trial to test the effects of dietary fiber, 120 healthy obese adolescents and young adults, age 12-21 (>97th percentile of BMI-for-age) will be recruited to participate in this study.

Recruitment outreach will begin with an email invitation. Parents will be encouraged to call a toll-free number for study information and answer via email. One email will be sent to potential study participants. If there is no response to the email, research staff will call parents up to 5 times and leave 3 messages to introduce the study. Once a parent or potential participant has been reached over the phone, research staff will explain the study and determine interest in participating. If member is interested in participating, research staff will email member the informed consent form (ICF). Participants will sign ICF using Adobe e-Sign web server.

Intervention: Participants will be instructed to consume 1 tea spoon of psyllium per day for 3 months and otherwise maintain their habitual diet. Using a mobile application, participants will be asked to track bowel movement and intestinal symptoms such as bloating and flatulence beginning two weeks prior to the intervention.

Liquid meal challenge test: The metabolic test will be conducted as two sessions lasting 180 minutes each, before and after the dietary fiber intervention (week 0 and 12). Subjects will participate in the metabolic tests after an overnight fast. Subjects will consume 250 ml of a standard liquid meal replacement shake with sugar added to 75 g of total sugar per meal (equivalent to oral glucose tolerance test used in clinical care). Blood draw will be done through an indwelling catheter in the antecubital vein and blood samples collected into 3 mL Ethylenediaminetetraacetic acid (EDTA) containing tubes at -15, 0, 30, 60, 90, 120, and 180 minutes after administration of the test meal. An additional 5 mL serum tube and urine will be collected at time -15 min. Total blood draw volume for the entire test is 26 mL.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Southern California (KPSC) member for at least 12 months.
* KPSC members ages 12 to 21 years old.
* KPSC member with >97th percentile of BMI for age.
* Minors with parents whose preferred language is English.
* 18 to 21 year old members whose preferred language is English.

Exclusion Criteria:

* Has diagnosis of serious mental illness and/or cognitive impairment.
* Provider has concerns over participation.
* Minors with parent whose preferred language is not English.
* 18 to 21 year old members whose preferred language is not English.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 3 year recruitment period
  Proportion of patients recruited/consented
Retention | 3-mo study period
  Proportion of participants remaining in study

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Clinical Research Center, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No